CLINICAL TRIAL: NCT04318197
Title: Personalized Rehabilitation Strategies According to Muscle Volume Before Knee Arthroplasty: a Pilot Study
Brief Title: Rehabilitation with Personalized Strategies According to Muscle Volume Before Knee Arthroplasty
Acronym: REPERAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lake of financing
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 29BRC.19.0154
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Gonarthrosis; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Global rehabilitation (Active Comparator): 2 hours of daily rehabilitation, 3 days per week during 4 weeks
  Interventions: Other: Global rehabilitation program
- Personalized rehabilitation (Experimental): 2 hours of daily rehabilitation including at least 2 times 20 minutes of electrostimulation on atrophied muscles, 3 days per week during 4 weeks
  Interventions: Other: Personalized rehabilitation program with electrostimulation
- Classic rehabilitation (No Intervention): 40 minutes of rehabilitation, once a week during 4 weeks.

INTERVENTIONS:
Other: Personalized rehabilitation program with electrostimulation — Patient with knee arthroplasty indication. After clinical assessment and a MRI measurement of muscle volume, patients start a 2 hours daily rehabilitation including 2 times 20 minutes of electrostimulation of atrophied muscles, 3 days per week during 4 weeks.
  Arms: Personalized rehabilitation
Other: Global rehabilitation program — Patient with knee arthroplasty indication. After clinical assessment and a MRI measurement of muscle volume, patient start a 2 hours daily rehabilitation targeting muscles groups with strengthening and stretching exercises, 3 days per week during 4 weeks.
  Arms: Global rehabilitation

SUMMARY:
Preoperative rehabilitation before total knee arthroplasty (TKA) has not been proven to be effective. Latest meta-analyzes do not find any improvement of motor performance during gait 6 months after surgery. However, most of the previous studies did not specifically target muscle atrophy to design rehabilitation protocol. Pre-operative muscle atrophy, although not systematic, is often observed. The preoperative muscles volumes of thigh muscles have been poorly identified and never used to adjust the pre operative rehabilitation strategy.

As part of the "FOLLOWKNEE" (RHU) project, which attempts to implement a personalized management of TKA and its follow-up, this study wants to explore the potential effect of adapted treatment to improve muscle force and muscle volume before TKA.

ELIGIBILITY:
Inclusion Criteria:

* Terminal stage gonarthrosis with total knee arthroplasty (TKA) indication
* TKA indicated by the surgeon
* Body Mass Index < 35
* Acceptance to realize a preoperative rehabilitation in outpatient setting
* Adult between 18 and 80 years old
* Patient affiliated to social security
* Patient who signed an informed consent

Exclusion Criteria:

* Functionally uncomfortable osteoarticular illness (disabling pain, functional limitation of joint amplitudes or muscle strength) of controlateral leg.
* Unable or refusal to consent
* Contraindication to electrostimulation (skin lesion, nearby implanted metallic material, implanted cardiac or neurologic electrostimulator, intolerance to muscle electrical stimulation)
* Unstable medical situation preventing the continuous realization of a program of at least 4 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Difference of isometric strength D0-W4p | Day 0 to Week 4 postoperative
  Isometric strength of quadriceps (QS) and hamstring (HS) will be measured on isokinetic bench and the difference between D0 and W4 will be calculated as follows : (QSW4p-QSD0)+(HSW4p-HSD0). Personalized rehabilitation will first be compared to classic rehabilitation and if positive to global rehabilitation.

SECONDARY OUTCOMES:
Difference of isometric strength D0-W4 | Day 0 to Week 4
  Isometric strength of quadriceps (QS) and hamstring (HS) will be measured on isokinetic bench and the difference between D0 and W4 (W4) will be calculated.
Difference of isometric strength D0-W12p | Day 0 to Week 12 postoperative
  Isometric strength of quadriceps (QS) and hamstring (HS) will be measured on isokinetic bench and the difference between D0 and W12postoperative (W12p) will be calculated.
Muscles volumes | Day 0, Week 4, Week 2 postoperative
  Quadriceps and hamstring volume as well as all muscles volume of each muscles groups will be evaluated in MRI.
Walking speed on 10 meters | Day 0, Week 4, Week 4 postoperative, Week 12 postoperative
  The patient will be timed when walking 10meters on a graduated corridor. They will be allowed to stop or use a technical help.
Time up and go test (TUG) | Day 0, Week 4, Week 4 postoperative, Week 12 postoperative
  The patient must get up from the sitting position and walk three meters from the chair and then retrace his steps (turn 180 degrees) and sit down again. The time that the person puts to this activity is timed by the evaluator.
Western Ontario McMaster Osteoarthritis Index (WOMAC) | Day 0, Week 4, Week 4 postoperative, Week 12 postoperative
  WOMAC is a medical scale for hip and osteoarthritic knee consisting of 24 questions scored between 0 and 4. The questions are about pain, joint stiffness and function.
Pain in Analogic Visual Scale (AVS) | Day 0, Week 4, Week 4 postoperative, Week 12 postoperative
  The pain during the 5 last days will be evaluated by Analogic Visual Scale. Pain is evaluated on a scale between 0 and 10. 0 is no pain and 10 the worse pain.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier REMY-NERIS, Pr, Principal Investigator — University hospital of Brest
Locations (1):
- CHRU de Brest, Brest, France, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement.